CLINICAL TRIAL: NCT03317795
Title: Prospective Randomized Trial of Tranexamic Acid Versus Levonorgestrel Intrauterine System for the Treatment of Heavy Menstrual Bleeding in Women With Uterine Fibroids
Brief Title: Treatment of Heavy Menstrual Bleeding in Women With Uterine Fibroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shannon K. Laughlin-Tommaso (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Shannon K. Laughlin-Tommaso, Associate Professor of Obstetrics and Gynecology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-008671; R21HD091337 (NIH)
Record Dates: First submitted 2017-10-10; First posted 2017-10-23 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Heavy Menstrual Bleeding; Menorrhagia; Uterine Fibroids
Keywords: Menorrhagia; FIbroids; Menstrual Bleeding; Heavy Bleeding; Menses; Uterine Fibroids
MeSH Terms: conditions — Menorrhagia; Leiomyoma | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levonorgestrel IUS (Active Comparator): Levonorgestrel-releasing intrauterine system (Mirena) contains 52 mg of levonorgestrel, a progestin, and is intended to provide an initial release of approximately 20 mcg/day. Levonorgestrel intrauterine system is effective immediately upon placement in the uterus and can be kept in place for up to 5 years.
  Interventions: Drug: Levonorgestrel IUS
- Tranexamic Acid (Active Comparator): Tranexamic Acid (Lysteda) is an antifibrinolytic drug. Tranexamic Acid will be dosed at 1300mg by mouth three times a day at the start of menses and used during the days that bleeding is heaviest (not to exceed 5 days per menstrual cycle).
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Levonorgestrel IUS — LNG-IUS was FDA-approved for the treatment of heavy menstrual bleeding in 2009 and previously for contraception in 2000. The LNG-IUS is a T-shaped device with a polyethylene body containing a hormone reservoir, holding a total of 52 mg of levonorgestrel. LNG-IUS initially releases 20 micrograms of the progestin per day, which decreases to less than half that amount after 5 years of use. The levonorgestrel causes stromal pseudodecidualization, decreases endometrial thickness, and lowers uterine vascular density.
  Other Names: Mirena IUS
  Arms: Levonorgestrel IUS
Drug: Tranexamic Acid — Tranexamic Acid was FDA-approved for the treatment of heavy menstrual bleeding in 2009. Tranexamic Acid is a plasminogen-activator inhibitor that blocks fibrinolysis and reduces plasmin activity. A special formulation was designed for the treatment of heavy menstrual bleeding that reduces gastrointestinal side effects, brand name Lysteda which will be prescribed as 1300 mg to be taken three times per day for up to 5 days of the menstrual period.
  Other Names: Lysteda
  Arms: Tranexamic Acid

SUMMARY:
This is a randomized controlled trial (RCT) to assess the comparative effectiveness of Levonorgestrel Intrauterine System (LNG-IUS) to Tranexamic Acid (TA) for the treatment of heavy menstrual bleeding (HMB) in women with clinically-significant fibroids.

DETAILED DESCRIPTION:
Uterine fibroids are common and debilitating problem for some women. Nearly 60% of women with fibroids report that symptoms affect their quality of life and impede physical activity, and 24% report that fibroid symptoms prevent them from reaching their true potential at work. Heavy menstrual bleeding, the most common symptom of uterine fibroids, affects approximately 1.4 million women per year.

Medical therapy is the first line treatment for heavy menstrual bleeding, but further studies need to be done to prove the effectiveness of these treatments.

The goal of this study is to determine the effectiveness of non-estrogenic medical therapy in women with a range of fibroid sizes, locations, and number.

Two effective medical treatments for heavy menstrual bleeding have limited data in women with fibroids. The Levonorgestrel intrauterine system was FDA approved for the treatment of heavy menstrual bleeding in 2009 and is highly effective for decreasing menstrual bleeding, treating anemia and improving quality of life. Moreover, it can be used continuously for 5 years. Tranexamic Acid is widely used outside the U.S. and was also FDA approved for heavy menstrual bleeding in 2009. Tranexamic Acid reduces menstrual blood loss in 40% of women and improves quality of life. In women with fibroids, Tranexamic Acid has been shown to decrease heavy menstrual bleeding and cause necrosis of the fibroids, especially larger fibroids, which should improve its efficacy for women with fibroids.

This randomized controlled trial will assess the comparative effectiveness of Levonorgestrel intrauterine system to Tranexamic Acid for the treatment of heavy menstrual bleeding in women with uterine fibroids

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women ages 25 -50
* Monthly menses
* Image-confirmed uterine fibroids of at least 1 cm in size, either submucosal or intramural
* Seeking treatment for heavy menstrual bleeding following completed clinical evaluation
* Self-reported heavy menstrual bleeding for three months or longer
* Completed evaluation for heavy menstrual bleeding within one year of study enrollment
* Understands the English language for consent and questionnaires
* Able and willing to provide informed consent

Exclusion Criteria:

* Class 0 fibroids confirmed by hysteroscopy, saline-infused sonogram, or 3D ultrasound
* Uterine sounding length ≥ 14 cm
* Uterine size ≥ 20 weeks gestational size
* Abnormal endometrial biopsy or incomplete clinical testing to rule out malignancy
* Needs or is using hormonal contraception, including estrogen-containing medications
* Venous thromboembolic history, clotting disorder, or strong family history of venous thromboembolic events
* Breast, uterine, or cervical malignancy
* Liver disease or liver tumor
* Pelvic inflammatory disease, gonorrhea or chlamydia infection during the past three months
* Hemoglobin < 8 mg/dL. For women with hemoglobin 8.0 - 12.0 mg/dL, iron supplement is recommended
* Serum creatinine ≥ 1.4
* Current pregnancy or currently lactating

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon K Laughlin-Tommaso, MD, MPH, Principal Investigator — Mayo Clinic; Christopher C Destephano, MD, MPH, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Jacksonville, Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Started | 9 | 9
Completed | 7 | 2
Not Completed | 2 | 7
Not completed — IUD Expulsion | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Treatment change | 0 | 3
Not completed — Intolerance of medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levonorgestrel IUS | Tranexamic Acid | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (5.6) | 44.7 (4.8) | 43.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 2
  White | 6 | 7 | 13
  Hispanic or Latino | 1 | 1 | 2
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Baseline hemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.1 (1.7) | 12.22 (1.9) | 12.2 (1.8)
Baseline ferritin [Median (Inter-Quartile Range); unit: mcg/L] | 6 [4 to 7] | 10 [5 to 56] | 7 [5 to 15]
Fibroid largest diameter [Median (Inter-Quartile Range); unit: cm] | 3.6 [2.3 to 5.2] | 2.5 [1.8 to 5.0] | 3.5 [2.0 to 5.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Reported Menorrhagia Scores
Description: The Menorrhagia Multi-Attribute Scale (MMAS) questionnaire captures the subjective consequences of menorrhagia on six domains: practical difficulties; social life; psychological wellbeing; physical health; work routine; and family life. Each of the six domains has four statements that represent four levels of response. Respondents indicate the statement that best matches their feelings for each domain. The statement scores derive from a weighting of the domains and a weighting of the statements in level of severity by women in the original study. Scores range from 0 (worst possible state in all domains) to 100 (best possible state in all domains).
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for 2 subjects in the Levonorgestrel IUS study arm and 3 subjects in the Tranexamic Acid study arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 7 | 6
score on a scale | 59.1 [34.1 to 63.7] | 25.4 [12.5 to 40.3]
Statistical Analysis 1: Comparison: Levonorgestrel IUS vs Tranexamic Acid; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Participants to Complete Study
Description: Total number of study participants to complete assigned treatment.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 9 | 9
Participants | 7 | 2

3. Secondary Outcome: Change in Pain Score
Description: Pain will be measured by a 10 cm visual analog scale (VAS) which uses a 100 point score, with 0 indicating no pain and 100 indicating worst pain ever. Change was determine by subtracting the 3 month score from baseline, a negative score indicates a decrease in pain.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 7 | 6
units on a scale | -57.5 [-60 to -30] | 0 [-63 to 20]
Statistical Analysis 1: Comparison: Levonorgestrel IUS vs Tranexamic Acid; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Quality of Life
Description: Measured by the RAND 36-Item Health Survey (Version 1.0). Physical function and mental well-being on scale range from 0-100. A high score defines a more favorable health state.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 7 | 6
units on a scale
  Physical Function | 11.1 [0.2 to 15.3] | 1.7 [-0.6 to 2.4]
  Mental Well-being | -1.0 [-9.1 to 11.6] | 3.3 [2.4 to 11.1]
Statistical Analysis 1: Comparison: Levonorgestrel IUS vs Tranexamic Acid; Physical composite score; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levonorgestrel IUS vs Tranexamic Acid; Mental composite score; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Quality of Life, as Measured by the Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL)
Description: The Uterine Fibroid Symptom and Health Related Quality of Life (HRQL) Questionnaire consists of an 8-item symptom severity scale and 29 HRQL items comprising 6 domains: Concern, Activities, Energy/Mood, Control, Self-consciousness, and Sexual Function. All items are scored on a 5-point Likert scale, ranging from "not at all" to "a very great deal" for symptom severity items and "none of the time" to "all of the time" for the HRQL items. Symptom severity and HRQL subscale scores are summed and transformed into a 0-100 point scale. Higher HRQL subscale scores indicate better HRQL.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 7 | 6
score on a scale | 32.8 [24.1 to 58.6] | 21.6 [10.3 to 39.7]
Statistical Analysis 1: Comparison: Levonorgestrel IUS vs Tranexamic Acid; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Symptoms, as Measured by the Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL)
Description: The Uterine Fibroid Symptom and Health Related Quality of Life (HRQL) Questionnaire consists of an 8-item symptom severity scale and 29 HRQL items comprising 6 domains: Concern, Activities, Energy/Mood, Control, Self-consciousness, and Sexual Function. All items are scored on a 5-point Likert scale, ranging from "not at all" to "a very great deal" for symptom severity items and "none of the time" to "all of the time" for the HRQL items. Symptom severity and HRQL subscale scores are summed and transformed into a 0-100 point scale. Higher Symptom Severity scores indicating greater symptoms.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 7 | 6
score on a scale | -28.1 [-37.5 to -21.9] | -15.6 [-21.9 to -3.1]
Statistical Analysis 1: Comparison: Levonorgestrel IUS vs Tranexamic Acid; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Fibroid Size
Description: Fibroid size will be reported as millimeters (mm).
Time Frame: 9 months
Population: Data not collected or analyzed for 1 subject in the Tranexamic Acid arm.
Measure: Median (Full Range); unit: mm
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
Number analyzed (Participants) | 7 | 1
mm | 3 [3 to 15] | 10.5 [3 to 18]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of 9 months on all participants.
Arm/Group | Levonorgestrel IUS | Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levonorgestrel IUS (N=9) | Tranexamic Acid (N=9)
Imbedded IUD (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Gastrointestinal Disturbance (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased Vaginal Bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03317795/Prot_SAP_000.pdf